CLINICAL TRIAL: NCT03965507
Title: A Cross-sectional Study of Patients, Who Diagnosed Lumbar Disc Hernia With or Without Sacroiliac Joint Dysfunction
Brief Title: The Prevalence Of Sacroiliac Joint Dysfunction In Patients With Lumbar Disc Hernia
Status: Completed | Type: Observational
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Hilal Telli, Assistant Professor - Medical Doctor, European University of Lefke
Other Study IDs: The Prevalence Of SJD
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Lumbar Disc Herniation; Sacroiliac Joint Dysfunction
Keywords: Disc hernia; Dysfunction; Lumbar; Sacroiliac joint
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Functional Residual Capacity; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group with sacroiliac joint dysfunction: The patient with sacroiliac joint dysfunction in lumbar disc hernia
  Interventions: Other: Evaluation of the prevalence of sacroiliac joint dysfunction in lumbar disc herniation
- The group without sacroiliac joint dysfunction: The patient without sacroiliac joint dysfunction in lumbar disc hernia
  Interventions: Other: Evaluation of the prevalence of sacroiliac joint dysfunction in lumbar disc herniation

INTERVENTIONS:
Other: Evaluation of the prevalence of sacroiliac joint dysfunction in lumbar disc herniation
  Other Names: Pain level; Presence of neuropathic pain; Functional capacity; Quality of life; Presence of depression; Presence of kinesiophobia

SUMMARY:
In this study evaluated the prevalence of sacroiliac joint dysfunction in patients with lumbar disc hernia and examined the variations in clinical parameters cause by this combination.

DETAILED DESCRIPTION:
Two hundred thirty-four patients already diagnosed with lumbar disc hernia were included in the study. During the evaluation, sacroiliac joint dysfunction was investigated using specific tests, pain levels with a Visual Analog Scale, and the presence of neuropathic pain using the Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale. Other clinical assessments were performed using the Beck Depression Inventory, Health Assessment Questionnaire, and Tampa Kinesiophobia Scale. Positivity in three out of six provocation tests was adopted as a criterion for sacroiliac joint dysfunction.

Sample Size A power analysis using the formula n= t2pq / d2 was performed to determine the sample size. Based on those data the investigators concluded that a minimum of 174 and a maximum of 322 patients would be required to achieve significant results, and 234 patients were enrolled.

Statistical Analysis The study data were expressed as mean plus standard deviation (SD) for constant variables values and as number and percentage for categoric variables. The chi-square test was used to analyze categoric variables. Results were evaluated at a 95% confidence interval at a significance level of p˂0.05. The analysis was performed on Statistical Package for the Social Sciences (SPSS) for Windows 16.0 software.

The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guideline has been implemented in this manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 - 60 years old
* Diagnosis of lumbar disc herniation
* To have sufficient cognitive level to fill clinical evaluation forms
* The patient agreed to participate in the study

Exclusion Criteria:

* Lumbar pain, the etiology of which was suspected to be inflammatory in character
* Structural vertebral deformity or fracture
* The severe and progressive neurological deficit
* A history of severe psychiatric disease
* Substance and/or alcohol dependence, with uncontrolled diabetes mellitus (DM), malignancy, spinal infection
* A history of vertebral surgery
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two hundred thirty-four patients already diagnosed with lumbar disc hernia were included in the study. 63.2% of patients were female and 36.8% were male. Mean age was 46.72 ± 11.14 years.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Evaluation the prevalence of sacroiliac joint dysfunction in patients with lumbar disc hernia | 1 day
  During the evaluation, sacroiliac joint dysfunction was investigated using specific tests. Positivity in three out of six provocation tests was adopted as a criterion for sacroiliac joint dysfunction.
Examination of the level of pain caused by this combination which with sacroiliac joint dysfunction in lumbar disc hernia | 1 day
  All patients were evaluated in terms of pain threshold measurements using a Visual Analogue Scale (VAS). The patient is asked to mark the severity of the pain on a horizontal or vertical 10 cm line. It is defined as 0 no pain, 5 moderate pain, 10 is the most severe pain encountered in life.
Examination the presence of depression caused by this combination which with sacroiliac joint dysfunction in lumbar disc hernia | 1 day
  The presence of depression was evaluated using the Beck Depression Inventory. The Beck Depression Inventory created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  Each answer is scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
  In this study evaluated that there is no depression between 0 and 13 points, a moderate depression of 14-24 points, and a severe depression of more than 25 points.
Effect on the quality of life this combination which with sacroiliac joint dysfunction in lumbar disc hernia: Health Assessment Questionnaire | 1 day
  Quality of life was performed using the Health Assessment Questionnaire.The Health Assessment Questionnaire (HAQ) was originally developed in 1978 by James F. Fries, MD, and colleagues at Stanford University. The domain of disability is assessed by the eight categories of dressing, arising, eating, walking, hygiene, reach, grip, and common activities. Discomfort is determined by the presence of pain and its severity. Each answer is rated 0-3. The Health Assessment Questionnaire (HAQ) is a questionnaire that reflects the functional status, and its score is correlated with disease activity indicators.
Examination the presence of kinesiophobia caused by this combination which with sacroiliac joint dysfunction in lumbar disc hernia | 1 day
  The presence of kinesiophobia was evaluated using the Tampa Kinesiophobia Scale.The Tampa Scale for Kinesiophobia (TSK)that was developed in 1990 is a 17 item questionnaire used to assess the subjective rating of Kinesiophobia or fear of movement. The original questionnaire was developed to "discriminate between non-excessive fear and phobia among patients with chronic musculoskeletal pain''. The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of Kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Telli, MD, Principal Investigator — European University of Lefke

IPD SHARING:
Plan to Share IPD: No
From an ethical point of view, this data should remain between the doctor and the patients. Therefore a plan is not created.

REFERENCES:
- [Background] van Tulder M, Malmivaara A, Esmail R, Koes B. Exercise therapy for low back pain: a systematic review within the framework of the cochrane collaboration back review group. Spine (Phila Pa 1976). 2000 Nov 1;25(21):2784-96. doi: 10.1097/00007632-200011010-00011. PMID 11064524
- [Result] Madani SP, Dadian M, Firouznia K, Alalawi S. Sacroiliac joint dysfunction in patients with herniated lumbar disc: a cross-sectional study. J Back Musculoskelet Rehabil. 2013;26(3):273-8. doi: 10.3233/BMR-130376. PMID 23893142
- [Result] Chou LH, Slipman CW, Bhagia SM, Tsaur L, Bhat AL, Isaac Z, Gilchrist R, El Abd OH, Lenrow DA. Inciting events initiating injection-proven sacroiliac joint syndrome. Pain Med. 2004 Mar;5(1):26-32. doi: 10.1111/j.1526-4637.2004.04009.x. PMID 14996234
- [Result] Prather H, Hunt D. Conservative management of low back pain, part I. Sacroiliac joint pain. Dis Mon. 2004 Dec;50(12):670-83. doi: 10.1016/j.disamonth.2004.12.004. No abstract available. PMID 15767995